CLINICAL TRIAL: NCT02154906
Title: Clinical and Radiographic Evaluation of Demineralized Freeze-Dried Bone Allograft Versus Platelet Rich Fibrin for the Treatment of Periodontal Intrabony Defects in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Brian L Mealey, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20130439H
Record Dates: First submitted 2014-05-29; First posted 2014-06-03 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Periodontitis
Keywords: periodontal disease; periodontitis
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFDBA (Active Comparator): DFDBA used to graft intrabony defect
  Interventions: Device: DFDBA
- autologous platelet rich fibrin (Experimental): autologous platelet rich fibrin used to graft intrabony defect
  Interventions: Device: autologous platelet rich fibrin

INTERVENTIONS:
Device: DFDBA
  Arms: DFDBA
Device: autologous platelet rich fibrin
  Arms: autologous platelet rich fibrin

SUMMARY:
Inflammatory periodontal disease often results in loss of bone around the teeth. Bone defects that have a certain size and shape (called intrabony or intraosseous defects) may be improved by using a graft material in the bony defect. The purpose of this study is to compare healing of periodontal intrabony defects that are treated using demineralized freeze dried bone allograft (DFDBA) versus autogenous platelet-rich fibrin.

The null hypotheses is that there will be no significant differences in bone fill, CAL gain, PD reduction or recession at sites treated with PRF compared to sites treated with DFDBA.

DETAILED DESCRIPTION:
This entire protocol involves procedures that are standard care. The purpose of the research is to evaluate whether there are any differences in results of periodontal surgical treatment using PRF in intrabony defects versus using DFDBA in intrabony defects. The DFDBA used in this study is an approved product and will be used in an approved manner. The PRF used in this study is an autologous product derived from the patient's own blood and is also being used in an approved manner during this study.

The primary outcomes evaluated in this study will include the soft tissue parameter of gain in clinical attachment level (CAL) and the hard tissue parameter of bone fill (BF). Secondary outcomes evaluated will include the soft tissue parameters of probing depth (PD) reduction and change in gingival recession (GR). These parameters will be evaluated over a 6-month period following intraoperative application of the material in advanced periodontal defects in 44 subjects (22 subjects per group with expected completion of 15 subjects per group). Six months after surgery, final post-operative clinical and radiographic measurements will be made.

Each subject will randomly be assigned (1:1) to receive either flap surgery with autologous platelet-rich fibrin (PRF) placed into the intrabony defect (test) or flap surgery with demineralized freeze-dried bone allograft (DFDBA) placed into the intrabony defect (control). Subjects will be randomized by drawing a sealed envelope from a stack of envelopes, each of which will contain a slip of paper on which is written PRF or DFDBA. The number of envelopes per group will equal the total number of subjects to be enrolled per group. Because collection and processing of PRF requires specific equipment, subjects will be randomized just prior to the surgical procedure being performed (before delivery of local anesthesia) rather than after flap reflection and debridement.

Each subject will contribute only 1 study site. If a subject has more than one interproximal bony defect in the area being treated surgically, only 1 such site will be chosen as the study site. The site with the deepest CEJ-BD measurement will be chosen. All other nonstudy sites in the surgical area will be treated with the same material as the adjacent study site (PRF or DFDBA). Clinical measurements at the time of surgery and at the 6-month follow-up will be made by one of two examiners who are masked as to study group. The same clinical examiner who makes measurements at the time of surgery will also make measurements at the 6-month follow-up.

Patients will be given post-operative antibiotics for 7 days after surgery as part of standard care (amoxicillin 500mg three times a day for 7 days; if allergic to amoxicillin, patients will receive doxycycline 100mg twice a day for 7 days). Subjects will be seen 10-14 days after surgery for routine follow-up procedures including removal of sutures and removal of visible plaque. Subjects will be followed again for routine postoperative procedures at 1 month, 2 months, and 4 months after surgery. The final postoperative visit will take place at 6 months post-surgery and will include final radiographic and clinical assessments of the study site. The study is over after this 6-month follow-up visit.

Routine radiographs will be made as standard care procedures pre-operatively and at the 6-month follow-up time point. Radiographs will be standardized using Rinn XCP holders with customized bite registrations, and a 1mm radiopaque square grid (Fixott-Everett grid) will be placed over digital sensor plates to allow ease of linear measurement on the digital radiographic images. Radiographic measurements will be made by a masked examiner. Hard tissue measurements made from the radiographs at baseline and 6-month follow-up will include CEJ to base of bony defect (CEJ-BD).Measurements will be made to the nearest 0.5mm.Bone fill is the linear change (in mm) in CEJ-BD measurement between baseline examination and 6-month follow-up.

Soft tissue measurements made at baseline and 6-month follow-up will include probing depth (PD = gingival margin to base of soft tissue pocket), clinical attachment level (CAL = CEJ to base of soft tissue pocket), and gingival recession (GR = CEJ to gingival margin) at each defect site. North Carolina 15mm (UNC-15) periodontal probes will be used and measurements will be rounded to the nearest 0.5mm.

Intraoperatively, the bony defect will be measured from CEJ-BD to the nearest 0.5mm. This measurement will be made from both the facial and lingual aspect of the interproximal defect (i.e., the depth of the interproximal bony defect will be measured from both the facial and lingual aspect to its deepest depth). In addition, the number of bony walls will be characterized into one of 7 categories: 1) 1-wall, 2) 2-wall, 3) 3-wall, 4) combination 1,2-wall defect, 5) combination 1,3-wall defect, 6) combination 2,3-wall, or 7) circumferential defects. At 6-month follow-up, clinical evaluation of bone fill will be made using transgingival probing in the periodontal pocket from the CEJ to the bony crest. This measurement will also be made from both the facial and lingual aspect of the interproximal defect. This standard care procedure is done using topical anesthetic. Surgical re-entry will not be performed.

For final analysis, the defect will be characterized at the location having the deepest CEJ-BD measurement at the time of surgery. For example, if treating a defect on the distal aspect of tooth #19 in which the CEJ-BD measurement is 8.5mm from the facial aspect and 7.5mm from the lingual at the time of surgery, changes in soft tissue parameters (CAL, PD, recession) and hard tissue parameters (bone fill) for that defect will be determined using PD, CAL, recession and bone fill measurements taken from the facial aspect only (rather than using the mean of facial and lingual measurements to characterize the defect).

ELIGIBILITY:
Inclusion Criteria:

* Patient currently a patient at dental school or eligible for treatment at dental school
* Patient resides within 50 mile radius of dental school and is eligible for treatment in Graduate Periodontics Clinic
* Diagnosis of chronic periodontitis with a treatment plan that includes surgical treatment of an intrabony defect adjacent to a natural tooth
* Willing and able to provide informed consent and be available for multiple follow-up visits for the duration of the study
* One or more sites with 1) a probing depth of 6mm or greater (>6mm), 2) a radiographic bony defect depth of greater than 3mm (>3mm), 3) sufficient keratinized tissue to allow complete coverage of the defect with gingival flaps, and 4) radiographic base of bony defect at least 2mm coronal to the apex of the tooth
* Female patients who have undergone a hysterectomy, tubal ligation or menopause, and non-pregnant women of child-bearing potential

Exclusion Criteria:

* not meeting inclusion criteria above
* Failure to attain adequate oral hygiene prior to surgery (minimum 80% plaque-free surfaces)
* History within the last 6 months of daily use of smokeless tobacco, pipe or cigar smoking, or cigarette smoking exceeding 10 cigarettes per day. Former smokers who quit more than 6 months before the study are eligible for enrollment. Current smokers who smoke less than 10 cigarettes per day are eligible for enrollment.
* Untreated acute or chronic infections in the region of the study site
* Tooth mobility of Grade 2 or higher at the tooth with the potential test site
* Clinical or radiographic signs of apical pathology, root fracture, untreated carious lesions on the root surface or at the CEJ, subgingival restorations on the tooth with the potential test site
* Sensitivity or allergy to Bacitracin, Gentamycin, Polymyxin B Sulfate, alcohol and/or surfactants

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health Science Center School of Dentistry, San Antonio, Texas, United States

REFERENCES:
- [Derived] Chadwick JK, Mills MP, Mealey BL. Clinical and Radiographic Evaluation of Demineralized Freeze-Dried Bone Allograft Versus Platelet-Rich Fibrin for the Treatment of Periodontal Intrabony Defects in Humans. J Periodontol. 2016 Nov;87(11):1253-1260. doi: 10.1902/jop.2016.160309. Epub 2016 Jun 28. PMID 27353441

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 subjects were enrolled but 3 withdrew prior to group assignment, leaving N=41 assigned to groups
Groups:
- DFDBA: DFDBA used to graft intrabony defect
  DFDBA
- Autologous Platelet Rich Fibrin: autologous platelet rich fibrin used to graft intrabony defect
  autologous platelet rich fibrin
Period: Overall Study
Arm/Group | DFDBA | Autologous Platelet Rich Fibrin
Started | 21 | 20
Completed | 19 | 17
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFDBA | Autologous Platelet Rich Fibrin | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Full Range); unit: years] | 52.3 [23 to 68] | 57.2 [38 to 73] | 55.0 [23 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36
Clinical Attachment Level [Mean (Full Range); unit: mm] | 6.7 [4 to 11] | 6.3 [4 to 8] | 6.5 [4 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: measurement of CAL at the time of surgical intervention will be compared with measurement of CAL and bone level 6 months after surgery
Time Frame: baseline and 6 months after surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DFDBA | Autologous Platelet Rich Fibrin
Number analyzed (Participants) | 19 | 17
mm | 1.21 (1.50) | 1.03 (0.86)

2. Secondary Outcome: Change in Radiographic Bone Level
Description: measurement of radiographic bone level at the time of surgical intervention will be compared with measurement of bone level 6 months after surgery
Time Frame: baseline and 6 months after surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DFDBA | Autologous Platelet Rich Fibrin
Number analyzed (Participants) | 19 | 17
mm | 1.14 (0.88) | 1.10 (1.01)

ADVERSE EVENTS:
Arm/Group | DFDBA | Autologous Platelet Rich Fibrin
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes